CLINICAL TRIAL: NCT02726386
Title: A Multicenter, International, Open-label, Safety Study of ND0612, a Solution of Levodopa/Carbidopa Delivered Via a Pump System as a Continuous Subcutaneous Infusion in Subjects With Advanced Parkinson's Disease
Brief Title: A Long Term Safety Study of ND0612 Administered as a Continuous SC Infusion in Advanced Parkinson's Disease
Acronym: BeyoND
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroDerm Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ND0612H-012
Record Dates: First submitted 2016-03-29; First posted 2016-04-01 (Estimated); Results first posted 2023-05-06 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 24-hour dosing regimen (Experimental): Continuous SC infusion over 24 hours: fixed day rate of up to 0.64 mL/h for 18 hours, followed by a night rate of 0.08 mL/h for 6 hours to deliver a total daily dose of up to 720/90 mg of levodopa/carbidopa.
  All patients who had been previously assigned to the 24-hour group in the prior study continued on this dosing regimen; patients who had previously been assigned to the 14-hour daytime regimen were switched to the 24-hour regimen.
  Interventions: Drug: ND0612
- 16-hour dosing regimen (Experimental): Continuous SC infusion for over 16 hours: fixed rate of 0.75 mL/h to deliver a total infusion dose of 720/90 mg of levodopa/carbidopa over 16 hours.
  The device is removed at night and patients in this group also receive a morning oral dose of levodopa/carbidopa upon awakening.
  Interventions: Drug: ND0612

INTERVENTIONS:
Drug: ND0612 — ND0612, a solution of levodopa/carbidopa (LD/CD) delivered continuously subcutaneously (SC) via an infusion pump system
  Other Names: ND0612H

SUMMARY:
This is a multi-center, international, open-label, safety study of ND0612, a solution of levodopa/carbidopa (LD/CD) delivered via a pump system as a continuous SC infusion in subjects with advanced Parkinson's Disease (PD).

DETAILED DESCRIPTION:
This is a multi-center, international, open-label, safety study of ND0612, a solution of LD/CD delivered via a pump system as a continuous SC infusion in subjects with advanced PD. Two cohorts of subjects are candidates for this study: subjects who completed treatment in study ND0612H-006 within one month prior to enrollment (Cohort 1) and ND0612 naïve subjects or subjects who completed treatment in a ND0612 clinical study more than one month before screening (Cohort 2). After screening procedures and confirmation of the inclusion/exclusion criteria, subjects and their study partners will be trained and assisted at their homes during the first week of treatment on the proper operation of the pump system. One mandatory home visit will be performed during the first week and then on a monthly basis during 12-months of treatment. Subjects will return for in-clinic visits at Week 1 and at Months 1, 2, 3, 4, 6, 9, and 12 for assessment of safety and efficacy variables. Subjects will be allowed to continue with study treatment for an optional treatment extension period of up to Month 102 and the clinic visits will be performed every 3 months to assess subject long-term safety. Safety follow-up visits will occur 1, 2, and 3 months after the last SC infusion of ND0612 or after early termination.

ELIGIBILITY:
INCLUSION CRITERIA:

Cohort 1.

1. Subject is able to, and has signed an Institutional Review Board/Ethics Committee (IRB/EC)-approved informed consent form (ICF).
2. Subject has completed the treatment period of study ND0612H-006 not more than one month prior to enrolling in ND0612H-012.
3. Willing and able to administer the SC infusion alone or with the assistance of a study partner and able to comply with the study specific procedures.

Cohort 2.

1. Male and female PD subjects of any race aged at least 30 years who sign an IRB/EC-approved ICF.
2. PD diagnosis consistent with the UK Brain Bank Criteria.
3. Modified Hoehn & Yahr scale in "ON" state of stage ≤3.
4. Taking at least 4 doses/day of LD/DDI (or at least 3 doses/day of Rytary) and taking, or have attempted to take, at least one other PD treatment for at least 30 days.
5. Subjects must be stable on their anti-PD medications for at least 30 days before Day 1.
6. Subjects may have had prior exposure to SC apomorphine injections/infusion but must have stopped continuous apomorphine administration at least 4 weeks before the screening visit. Treatment with apomorphine is prohibited during the entire ND0612 treatment period.
7. Must have a minimum of 2 hrs of "OFF" time per day with predictable early morning "OFF" periods as estimated by the subject.
8. Must have predictable and well defined early morning "OFF" periods with a good response to LD for treatment of the early morning "OFF" in the judgement of the investigator.
9. Mini Mental State Examination (MMSE) score ≥26.
10. No clinically significant medical, psychiatric or laboratory abnormalities which the investigator judges would be unsafe or non-compliant in the study.
11. Female subjects must be surgically sterile (hysterectomy, bilateral oophorectomy, or tubal ligation), postmenopausal (defined as cessation of menses for at least 1 year), or willing to practice a highly effective method of contraception. All female participants must be non-lactating and non-pregnant and have a negative urine pregnancy test at Screening and at Baseline. Female subjects of childbearing potential must practice a highly effective method of contraception (e.g., oral contraceptives, intrauterine devices, partner with vasectomy), 1 month before enrollment, for the duration of the study, and 3 months after the last dose of study drug. Alternatively, true abstinence is acceptable when it is in line with the subject's preferred and usual lifestyle. If a subject is usually not sexually active but becomes active, the subject and sexual partner must comply with the contraceptive requirements detailed above.
12. Willing and able to administer the SC infusion alone or with the assistance of a study partner after a screening period of up to 40 days and willing and able to comply with study requirements.
13. Subjects should have a named study partner.

EXCLUSION CRITERIA:

Cohort 1 and 2. Previously unable to tolerate ND0612 and/or have experienced intolerable adverse drug reactions associated with its use, regardless of the dosing regimen administered.

Cohort 2.

1. Atypical or secondary parkinsonism.
2. Acute psychosis or hallucinations in past 6 months.
3. Any relevant medical, surgical, or psychiatric condition, laboratory value, or concomitant medication which, in the opinion of the Investigator makes the subject unsuitable for study entry or potentially unable to complete all aspects of the study.
4. Any malignancy in the 5 years prior to randomization (excluding basal cell carcinoma of the skin or cervical carcinoma in situ that have been successfully treated).
5. Positive serum serology for Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) or Human Immunodeficiency Virus (HIV) at the Screening visit.
6. Prior neurosurgical procedure for PD, or Duodopa treatment
7. Subjects with a history of drug abuse or alcoholism within the past 12 months.
8. Clinically significant ECG rhythm abnormalities.
9. Renal or liver dysfunction that may alter drug metabolism including: serum creatinine >1.3 mg/dL, serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2 x upper limit of normal (ULN), total serum bilirubin >2.5 mg/dL.
10. Current participation in a clinical trial with an investigational product or past participation within the last 30 days before Day 1.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2027-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Salin, MD, Study Director — NeuroDerm Ltd.
Locations (57):
- United States (26):
  - Xenoscience, Phoenix, Arizona
  - Clinical Trials Inc., Little Rock, Arkansas
  - The Parkinsons and Movement Disorder Institute, Fountain Valley, California
  - Neuro Pain Medical Center, Fresno, California
  - University of Colorado Denver, Aurora, Colorado
  - Rocky Mountain Movement Disorders Center, Englewood, Colorado
  - Parkinson's Disease and Movement Disorder Center of Boca Raton, Boca Raton, Florida
  - MD Clinical, Hallandale, Florida
  - Infinity Clinical Research, LLC, Hollywood, Florida
  - University of Florida Health at Jacksonville, Jacksonville, Florida
  - Neurology Associates, PA, Maitland, Florida
  - Parkinsons Disease Treatment Center of Southwest Florida, Port Charlotte, Florida
  - Suncoast Neuroscience Associates, St. Petersburg, Florida
  - Infinity Clinical Research, LLC, Sunrise, Florida
  - USF Health Parkinson's Disease and Movement Disorders, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Unity Point Health, Des Moines, Iowa
  - University of Maryland, Neurology, Baltimore, Maryland
  - QUEST Research Institute, Farmington Hills, Michigan
  - Henry Ford Hospital, West Bloomfield, Michigan
  - Pyramid Clinical Research, Somerset, New Jersey
  - University of Cincinnati, Cincinnati, Ohio
  - The Movement Disorder Clinic of Oklahoma, Tulsa, Oklahoma
  - Synergy Trials, Richmond, Virginia
  - Sentara Neuroscience Institute, Virginia Beach, Virginia
  - Premier Research, Spokane, Washington
- Medical University Innsbruck, Innsbruck, Austria
- Czechia (3):
  - NEUROHK, s.r.o., Choceň
  - Clintrial s.r.o., Prague
  - Vestra Clinics, s.r.o., Rychnov nad Kněžnou
- France (7):
  - Centre Hospitalier d'Aix, Aix-en-Provence
  - CHU d'Amiens, Hopital Sud, Amiens
  - Hopital Neurologique Pierre Wertheimer, Bron
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Hopital Roger Salengro, Lille
  - Hopital de la Timone, Marseille
  - CHU de Poitiers, Poitiers
- Germany (6):
  - Kliniken Beelitz GmbH, Beelitz-Heilstätten
  - St. Josefs Hospital, Bochum
  - Klinikum-Bremerhaven Reinkenheide, Bremerhaven
  - Universitaetsklinikum Carl Gustav Carus an der Technischen Universitaet Dresden, Dresden
  - Klinik Haag, Haag in Oberbayern
  - Universitaets-und Rehabilitationskliniken Ulm, Ulm
- Israel (5):
  - Barzilai MC, Ashkelon
  - Hadassah Medical Center, Ein-Kerem Campus, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
- Italy (4):
  - University Foundation, Chieti
  - AOU Pisa, Pisa
  - IRCCS San Raffaele Pisana, Rome
  - IRCCS Hospital San Camillo Venice, Venice
- Poland (3):
  - Centrum Medyczne PLEJADY, Krakow
  - Krakowska Akademia Neurologii Sp. z o.o., Krakow
  - Indywidualna Praktyka Lekarska prof. dr hab, Lublin
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de la Princesa, Madrid

REFERENCES:
- [Result] Poewe W, Stocchi F, Arkadir D, Ebersbach G, Ellenbogen AL, Giladi N, Isaacson SH, Kieburtz K, LeWitt P, Olanow CW, Simuni T, Thomas A, Zlotogorski A, Adar L, Case R, Oren S, Fuchs Orenbach S, Rosenfeld O, Sasson N, Yardeni T, Espay AJ; BeyoND study group. Subcutaneous Levodopa Infusion for Parkinson's Disease: 1-Year Data from the Open-Label BeyoND Study. Mov Disord. 2021 Nov;36(11):2687-2692. doi: 10.1002/mds.28758. Epub 2021 Sep 8. PMID 34496081

RESULTS

PARTICIPANT FLOW:
Groups:
- 24-hour Dosing Regimen: Continuous SC infusion over 24 hours: fixed day rate of up to 0.64 mL/h for 18 hours, followed by a night rate of 0.08 mL/h for 6 hours to deliver a total daily dose of up to 720/90 mg of levodopa/carbidopa.
  All patients who had been previously assigned to the 24-hour group in the prior study continued on this dosing regimen; patients who had previously been assigned to the 14-hour daytime regimen were switched to the 24-hour regimen.
  ND0612: ND0612, a solution of levodopa/carbidopa (LD/CD) delivered continuously subcutaneously (SC) via an infusion pump system
- 16-hour Dosing Regimen: Continuous SC infusion for over 16 hours: fixed rate of 0.75 mL/h to deliver a total infusion dose of 720/90 mg of levodopa/carbidopa over 16 hours.
  The device is removed at night and patients in this group also receive a morning oral dose of levodopa/carbidopa upon awakening.
  ND0612: ND0612, a solution of levodopa/carbidopa (LD/CD) delivered continuously subcutaneously (SC) via an infusion pump system
Period: Overall Study
Arm/Group | 24-hour Dosing Regimen | 16-hour Dosing Regimen
Started | 90 | 124
Completed | 52 | 68
Not Completed | 38 | 56
Not completed — Adverse Event | 17 | 20
Not completed — Withdrawal by Subject | 14 | 28
Not completed — Other reasons | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 24-hour Dosing Regimen | 16-hour Dosing Regimen | Total
Number analyzed (Participants) | 90 | 124 | 214
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (8.9) | 63.9 (8.9) | 64.0 (8.9)
Age, Customized [Count of Participants; unit: Participants]
  Age (years): <65 years | 43 | 63 | 106
  Age (years): ≥65 years | 47 | 61 | 108
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 40 | 72
  Male | 58 | 84 | 142
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Caucasian | 86 | 116 | 202
  Ethnicity: Other | 4 | 8 | 12
BMI [Mean (Standard Deviation); unit: kg/m^2] — BMI = Body mass index
  kg/m^2 | 27.0 (5.5) | 27.2 (5.9) | 27.1 (5.7)
BMI [Count of Participants; unit: Participants]
  <20 kg/m2 | 11 | 11 | 22
  ≥20 kg/m2 | 79 | 113 | 192
Modified Hoehn & Yahr [Count of Participants; unit: Participants] — MODIFIED HOEHN AND YAHR STAGING:
  Stage 0 = No signs of disease. Stage 1 = Unilateral disease. Stage 1.5 = Unilateral plus axial involvement. Stage 2 = Bilateral disease, without impairment of balance. Stage 2.5 = Mild bilateral disease, with recovery on pull test. Stage 3 = Mild to moderate bilateral disease; some postural instability; physically independent.
  Stage 4 = Severe disability; still able to walk or stand unassisted. STAGE 5 = Wheelchair bound or bedridden unless aided.
  Participants
    <2 | 4 | 5 | 9
    2 | 37 | 52 | 89
    2.5 | 17 | 32 | 49
    3 | 32 | 35 | 67
MMSE total score [Mean (Standard Deviation); unit: Points] — Mini-Mental State examination (MMSE) is a 30-point questionnaire that is used to measure cognitive impairment. The range of the MMSE total score is from 0 to 30 points. Any score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment. The MMSE examination is performed at Screening in order to ensure that only patients with normal cognition are enrolled in the study (i.e. score of 24 points or more).
  Points | 28.8 (1.2) | 28.8 (1.2) | 28.8 (1.2)
Time since PD diagnosis [Mean (Standard Deviation); unit: years] | 10.6 (5.3) | 7.9 (3.8) | 9.0 (4.7)
Time since onset of fluctuations [Mean (Standard Deviation); unit: years] | 5.3 (4.3) | 5.2 (4.2) | 5.3 (4.2)
Total daily levodopa dose [Mean (Standard Deviation); unit: mg] | 1090 (623) | 1004 (540) | 1040 (577)
Total daily levodopa frequency [Mean (Standard Deviation); unit: Times per day] | 5.9 (2.2) | 5.1 (1.7) | 5.5 (2.0)
Concomitant medications [Count of Participants; unit: Participants]
  Dopamine agonists | 52 | 58 | 110
  MAO-B inhibitors | 37 | 44 | 81
  COMT inhibitors | 28 | 24 | 52
  Amantadine | 25 | 30 | 55

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events (Long-term Safety)
Description: Long-term safety (systemic and local) assessment will be based on adverse events (AEs), with a focus on adverse events of special interest (AESI), i.e., infusion site reactions, cases of hypersensitivity, polyneuropathy.
Time Frame: Baseline to Month 12
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | 24-hour Dosing Regimen | 16-hour Dosing Regimen
Number analyzed (Participants) | 90 | 124
Participants
  Any TEAE | 78 | 105
  Drug-related TEAEs | 65 | 78
  Infusion site TEAEs | 55 | 66
  Serious TEAEs | 17 | 14
  Death | 0 | 1

2. Primary Outcome: Percentages of Subjects Who Complete the 12-month Treatment Period or Discontinue Due to AE (Tolerability)
Description: Tolerability will be assessed based on the percentage of subjects that complete the 12-month treatment period of the study and the percentage of subjects who discontinue from the 12-month treatment period due to an AE.
Time Frame: Baseline to Month 12
Population: Intention-to-Treat (ITT) set
Measure: Count of Participants; unit: Participants
Arm/Group | 24-hour Dosing Regimen | 16-hour Dosing Regimen
Number analyzed (Participants) | 90 | 124
Participants
  Completed the 12-month treatment period | 52 | 68
  Discontinued due to AE | 17 | 20

3. Secondary Outcome: Adverse Events (Long-term Safety)
Description: Long-term safety (systemic and local) and tolerability will be based on AEs, with a focus on AESI, i.e., infusion site reactions, cases of hypersensitivity, polyneuropathy.
Time Frame: Month 12 to Month 102
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Change of Daily "ON" Time Without Troublesome Dyskinesia
Description: Exploratory endpoint. "ON" time without troublesome dyskinesia is defined as the sum of "ON" time without dyskinesia and "ON" time with non-troublesome dyskinesia. Daily "ON" time without troublesome dyskinesia will be assessed based on home "ON/OFF" diaries and normalized to 16 hours of awake time.
Time Frame: Baseline to Month 12
Reporting Status: Not Posted, anticipated posting 2028-02

5. Other Pre Specified Outcome: Change of Daily "OFF" Time
Description: Exploratory endpoint. Daily "OFF" time will be assessed based on home "ON/OFF" diaries and normalized to 16 hours of awake time.
Time Frame: Baseline to Month 12
Reporting Status: Not Posted, anticipated posting 2028-02

6. Other Pre Specified Outcome: Change of Total Daily Dose of Oral LD/DDI
Description: Exploratory endpoint. Total daily dose of oral Levodopa (LD)/Dopa-Decarboxylase Inhibitor (DDI).
Time Frame: Baseline to Month 12
Reporting Status: Not Posted, anticipated posting 2028-02

7. Other Pre Specified Outcome: Proportion of Responders
Description: Exploratory endpoint. A responder is defined as a subject that experiences ≥50% reduction in "OFF" time from Baseline. Improvement of ≥50% in "OFF" time will be assessed based on home "ON/OFF" diaries and normalized to 16 hours of awake time.
Time Frame: Baseline to Month 12
Reporting Status: Not Posted, anticipated posting 2028-02

8. Other Pre Specified Outcome: Change of Daily "ON" Time With Troublesome Dyskinesia
Description: Exploratory endpoint. Daily "ON" time with troublesome dyskinesia will be assessed based on home "ON/OFF" diaries in a subset of subjects who had more than 1 hour of troublesome dyskinesia at baseline. It will be normalized to 16 hours of awake time.
Time Frame: Baseline to Month 12
Reporting Status: Not Posted, anticipated posting 2028-02

9. Other Pre Specified Outcome: Change of PDQ-39 Scores
Description: Exploratory endpoint. Quality of Life in Parkinson's Disease (PDQ)-39 is a 39-item, self-administered questionnaire with 8 discrete dimensions (mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort.). The PDQ-39 Summary Index is the sum of the dimension scores divided by the number of dimensions. Higher scores indicate a worse quality of life.
Time Frame: Baseline to Month 12
Reporting Status: Not Posted, anticipated posting 2028-02

10. Other Pre Specified Outcome: Change of EQ-5D-5L Scores
Description: Exploratory endpoint. The perception of general quality of life (QoL) will be rated by the subjects using the EuroQoL 5-dimensions 5-severity levels (EQ-5D-5L) questionnaire. The EQ-5D-5L consists of 2 pages, the EQ-5D-5L descriptive system and the EQ Visual Analogue Scale (VAS). The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The EQ VAS records the respondent's self-rated health on a 20 cm vertical VAS with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'. Decrease in the 5-dimensions scores and increase in EQ VAS score will indicate improvement.
Time Frame: Baseline to Month 12
Reporting Status: Not Posted, anticipated posting 2028-02

11. Other Pre Specified Outcome: Change of UPDRS Part II (ADL)
Description: Exploratory endpoint. The Unified Parkinson's disease rating scale (UPDRS) is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The UPDRS Part II (activity of daily living) score was calculated as the sum of the individual UPDRS items 5-17. The Part II score is the sum of the answers to the 13 questions that comprise Part II, each of which are measured on a 5-point scale (i.e., 0 is normal and 4 indicates a severe abnormality). Higher scores correlate with greater impairments for daily activities.
Time Frame: Baseline to Month 12
Reporting Status: Not Posted, anticipated posting 2028-02

12. Other Pre Specified Outcome: Change in CGI-Severity and CGI-Improvement
Description: Exploratory endpoint. Clinical Global Impression (CGI) Severity (CGI-S) and Improvement (CGI-I) are rated by the investigator or designee. CGI-S employs a 7-point scale with 1 being "not at all ill" and 7 being "among the most severely ill subjects" for severity rating. The CGI-I employs a 7-point scale with 1 being "very much improved" and 7 being "very much worse" for improvement rating.
Time Frame: Baseline to Month 12
Reporting Status: Not Posted, anticipated posting 2028-02

13. Other Pre Specified Outcome: Change in SGI-Improvement
Description: Exploratory endpoint. Subjects Global Impression of Improvement (SGI-I) is rated by the subject. The SGI-I employs a 7-point scale with 1 being "very much improved" and 7 being "very much worse" for improvement rating.
Time Frame: Baseline to Month 12
Reporting Status: Not Posted, anticipated posting 2028-02

14. Other Pre Specified Outcome: Change in PDSS-2 Total Score
Description: Exploratory endpoint. The quality of night sleep is rated by the subjects using the Parkinson's Disease Sleep Scale (PDSS)-2, which includes questions addressing 15 commonly reported symptoms associated with sleep disturbance in PD. Higher scores indicate a lower quality of sleep, i.e., a reduction in the score indicates an improvement in sleep quality.
Time Frame: Baseline to Month 12
Reporting Status: Not Posted, anticipated posting 2028-02

15. Other Pre Specified Outcome: Change in UPDRS Part III (Motor Score)
Description: Exploratory endpoint. The Unified Parkinson's Disease Rating Scale (UPDRS) is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. UPDRS part III (motor) score is calculated as the sum of the individual UPDRS items 18-31, each of which are measured on a 5-point scale (i.e., 0 is normal and 4 indicates a severe abnormality). Higher scores correlate with greater motor impairment.
Time Frame: Baseline to Month 12
Reporting Status: Not Posted, anticipated posting 2028-02

16. Other Pre Specified Outcome: Change in Percentage of "OFF" Time and Percentage of Good "ON" During the First 3 Hours Since the Subject is Awake After 06:00 (6 am)
Description: Exploratory endpoint. Good "ON" time (or "ON" time without troublesome dyskinesia) is defined as the sum of "ON" time without dyskinesia and "ON" time with non-troublesome dyskinesia. For this endpoint, Good "ON" time and "OFF" time will be assessed based on home "ON/OFF" diaries during the first 3 hours since the subject is awake after 06:00 (6 am).
Time Frame: Baseline to Month 12
Reporting Status: Not Posted, anticipated posting 2028-02

17. Other Pre Specified Outcome: Change in ND0612 Total Dose
Description: Exploratory endpoint. Change in ND0612 total daily dose.
Time Frame: Baseline to Month 12
Reporting Status: Not Posted, anticipated posting 2028-02

18. Other Pre Specified Outcome: Proportion of Patients Who Reduced ND0612 Total Dose
Description: Exploratory endpoint. Proportion of patients who reduced ND0612 total dose at any time during the study.
Time Frame: Baseline to Month 102
Reporting Status: Not Posted, anticipated posting 2028-02

ADVERSE EVENTS:
Time Frame: Baseline to Month 12
Description: TEAEs are defined as all AEs that started or worsened on or after the start of first study drug administration or within 28 days after the last study drug administration in the present study and up to 12 months.
Arm/Group | 24-hour Dosing Regimen | 16-hour Dosing Regimen
All-Cause Mortality (participants affected / at risk) | 0/90 | 1/124
Serious Adverse Events (participants affected / at risk) | 17/90 | 14/124
Other Adverse Events (participants affected / at risk) | 69/90 | 82/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 24-hour Dosing Regimen (N=90) | 16-hour Dosing Regimen (N=124)
Cardiac disorder (Cardiac disorders) | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Infusion Site Hematoma (General disorders) | 1 | 0
Infusion site dermatitis (General disorders) | 0 | 1
Infusion site infection (General disorders) | 3 | 2 — Group term
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute polyneuropathy (Nervous system disorders) | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 1
Dystonia (Nervous system disorders) | 0 | 1
Hyperkinesia (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
On and off phenomenon (Nervous system disorders) | 2 | 1
Parkinsonism hyperpyrexia syndrome (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 1 | 0
Delusion (Psychiatric disorders) | 0 | 1
Impulse-control disorder (Psychiatric disorders) | 1 | 0
Paranoia (Psychiatric disorders) | 0 | 1
Paranasal sinus haematoma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Gastrointestinal tube insertion (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 24-hour Dosing Regimen (N=90) | 16-hour Dosing Regimen (N=124)
Nausea (Gastrointestinal disorders) | 3 | 15
Fatigue (General disorders) | 0 | 7
Infusion site edema (General disorders) | 5 | 5
Infusion site erythema (General disorders) | 9 | 7
Infusion site eschar (General disorders) | 2 | 15
Infusion site hematoma (General disorders) | 24 | 30
Infusion site infection (General disorders) | 13 | 9
Infusion site nodule (General disorders) | 31 | 35
Infusion site pain (General disorders) | 13 | 15
Urinary tract infection (Infections and infestations) | 7 | 12
Fall (Injury, poisoning and procedural complications) | 12 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Dyskinesia (Nervous system disorders) | 8 | 7
Anxiety (Psychiatric disorders) | 2 | 8
Depression (Psychiatric disorders) | 1 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review and approve any results of the study or abstracts for professional meetings prepared by the investigator(s). Published data must not compromise the objectives of the study. Data from individual study centers in multicenter studies must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2020-12-28): https://cdn.clinicaltrials.gov/large-docs/86/NCT02726386/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/86/NCT02726386/SAP_001.pdf